CLINICAL TRIAL: NCT05213988
Title: Effects on GLUcose Homeostasis of Changes in Plasma Lipoproteins Induced by Nutritional and Pharmacologic STrategies Against Diabetes-Related Metabolic Diseases
Brief Title: Effects on Glucose Homeostasis of Changes in Plasma Lipoproteins Induced by Nutritional and Pharmacologic Strategies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Andrea Natali, Full Professor, Azienda Ospedaliero, Universitaria Pisana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: GLUCO-STAR
Record Dates: First submitted 2021-12-06; First posted 2022-01-28 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Glucose Metabolism Disorders
MeSH Terms: conditions — Glucose Metabolism Disorders | interventions — Fibric Acids; Diet, High-Protein Low-Carbohydrate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low-Carbohydrate/High-Protein Diet (Experimental)
  Interventions: Dietary Supplement: Low-Carbohydrate/High-Protein diet
- Fibrate (Experimental)
  Interventions: Drug: Fibrates
- Intermittent Fasting (Experimental)
  Interventions: Dietary Supplement: Intermittent Fasting
- Control (No Intervention)

INTERVENTIONS:
Dietary Supplement: Intermittent Fasting — Intermittent fasting meal pattern
  Arms: Intermittent Fasting
Drug: Fibrates — Bezafibrate 400 mg/day
  Arms: Fibrate
Dietary Supplement: Low-Carbohydrate/High-Protein diet — Low-calorie, low-carbohydrate, high-protein diet
  Arms: Low-Carbohydrate/High-Protein Diet

SUMMARY:
The investigators aim to examine the impact of changes in plasma lipoproteins induced by nutritional and pharmacological interventions on glucose homeostasis

ELIGIBILITY:
Inclusion Criteria:

* age 18-65 years
* both males and females

Exclusion Criteria:

* acute or chronic conditions influencing glucose and lipid metabolism
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-07-30 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Glucose tolerance | 180 minutes
  Glucose tolerance will be measured as the area under the curve of plasma glucose levels in response to a 180-minute 75g oral glucose tolerance test (OGTT)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Natali, MD, Principal Investigator — University of Pisa
Locations (1):
- Azienda Ospedaliero-Universitaria Pisana, Pisa, PI, Italy

IPD SHARING:
Plan to Share IPD: No